CLINICAL TRIAL: NCT01727219
Title: COPD Assessment Test Can Predict Depression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-I010
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2011-02

CONDITIONS: Depression,; COPD
MeSH Terms: conditions — Depression; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The frequency of depression in COPD patients are substantial and early detection and prevention of depression is critical.

Recently, COPD assessment test (CAT) was developed and validated to assess the impact of COPD on patients' quality of life.

In this prospective study, we will investigate the predictive utility of CAT for predicting depression in COPD patients.

DETAILED DESCRIPTION:
This study is aimed to investigate the association between the COPD Assessment Test (CAT) and depression in stable COPD patients. Stable COPD patients will be enrolled from the tertiary hospitals. All patients will undergo lung function tests. The Korean versions of the CAT (COPD assessment test) and Patient Health Questionnaire-9 (PHQ-9) will be used to assess COPD symptoms and depressive disorder, respectively.

We will compare the depresssion frequency among GOLD classifications of airway limitation and among the four CAT groups. And. we will also investigate which items of the CAT are the strongest indicators of depression.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients who aged > or = 40 years

Exclusion Criteria:

* acute exacerbation within 3 months
* bronchial asthma or an increase in FEV1 of more than 12% of the predicted value with the use of 400 µg of albuterol.
* other lung diseases such as bronchiectasis, interstitial lung disease, and tuberculosis-destroyed lungs.
* who denied to consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable COPD patients who visit outpatient departments.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-02 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
The predictive utility of the COPD assessment test (CAT) scores for predicting depression in COPD patients | 1 year
  The association of CAT with depression score

CONTACTS AND LOCATIONS:
Overall Officials: KI-Suck Jung, Dr., Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Department of Pulmonary, Critical Care Medicine, Anyang-si, Gyeonggi-do, South Korea